CLINICAL TRIAL: NCT05165537
Title: Evaluation of Novel and Adapted MR Spectroscopy and Metabolic Imaging Techniques for Non-invasive Monitoring of Metabolite Levels in Humans in Physiologic States of Everyday Life
Brief Title: Non-Invasive Monitoring Of Metabolite Levels Using Novel And Adapted MR Spectroscopy Techniques
Acronym: NIMM_MRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NIMM_MRS
Record Dates: First submitted 2021-12-07; First posted 2021-12-21 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Magnetic Resonance Spectroscopy
Keywords: brain; muscle; healthy subjects; precision; repeatability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIMM_MRS (Experimental): testing of new MRS methods
  Interventions: Device: NIMM_MRS

INTERVENTIONS:
Device: NIMM_MRS — evaluation of new MRS methods

SUMMARY:
This Swiss National Science Foundation (SNF) funded project and the linked European project aim

* to improve magnetic resonance (MR) methods, specifically MR spectroscopy and metabolic imaging (making them more sensitive and accurate - also less dependent on motion),
* to extend them (making previously unobservable metabolites visible) and also
* to make them more stable (suitable for routine clinical use).

Magnetic resonance spectroscopy (MRS) is closely related to the widely used magnetic resonance imaging (MRI). Both methods are based on the same physical effect and are performed on the same equipment. However, while MRI mainly images the anatomy inside the body, MRS gives us information about the metabolism of the tissue. The main goal of this study is to develop and improve methods of MRS to better measure the concentrations of endogenous substances without actual intervention. MRS methodology development is performed in 4 steps:

1. A new method is developed and optimized theoretically and in sample preparations (solutions of chemicals).
2. The new methodology is evaluated in single healthy volunteers and optimized step by step for the conditions of use in the human body.
3. The methodology in evaluated in small groups of healthy volunteers (measurement accuracy and range of variation in healthy volunteers).
4. Feasibility is studied in different situations with possibly different metabolic situations (e.g. awake versus asleep or before and after muscular exertion).

For this purpose, about 100 subjects will be measured for different subprojects. Thus, among other things, one determines the measurement accuracy and also normal values in healthy subjects for the assessment of diseases in future studies.

DETAILED DESCRIPTION:
Magnetic resonance imaging (MRI) and spectroscopy (MRS) provide non-invasive modalities to explore human morphology, function and metabolism. MRS methods are in widespread use in clinical research and to some degree in clinical applications. MRS methodology has been continuously extended for the last 30 years. All extensions employing novel MR pulse sequences (acquisition software), acquisition hardware capabilities of MRI scanners or post-processing methods have to be validated in theory, and in practice, where they are first tested in vitro and then in healthy subjects. The proposed project is based on a SNF project and a Horizon 2020 project of the sponsor-investigator, where multiple methodological extensions of MRS sequences are implemented for improved measurements of metabolite levels, characteristics and maps.

The intended study uses MRI-scanners which have a Conformité Européenne (CE) label for diagnostic use. The manufacturer of the MR scanner provides a "research-license mode" with the very same hardware; however, since the flexibility of this mode of operation makes a CE process prohibitively long and complex, no CE label was aimed at for the research-license mode.

The methodological developments within the proposed study aim at novel or improved sequences, which have the potential to observe previously undetectable metabolites and to evaluate metabolite changes as function of time-of-day or previous exercise. The sequences are applied in investigations of healthy adult subjects in everyday physiological situations to document the potential of the novel methods in terms of accuracy, precision, robustness. Without such investigations on healthy subjects the methodological advances cannot be verified in a valid situation and thus not ported to more specific research trials or clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* healthy (no neuronal or metabolic diseases as stated by the study participant)
* able to lie still in the MR scanner for at least one hour

Exclusion Criteria:

* <18 yrs of age
* pregnancy or current state of lactation
* active implants
* passive ferromagnetic implants
* passive non-ferromagnetic metallic implants > 4 cm inside a region covered by the active radio-frequency (RF) coils
* large tattoos inside a region covered by the active RF coils
* known or suspected non-compliance,
* under-weight (<35 kg body weight)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
healthy-cohort signal intensity characteristics for metabolites of interest (MOI) | 2 months
  healthy-cohort signal intensity characteristics for MOI as targeted by newly developed/optimized MRS sequences. Novel MRS sequences will be administered in a small cohort of healthy subjects and each sequence will provide detection/quantification of one or multiple specific metabolites (or metabolite characteristics (e.g. diffusivity)). Respective cohort averages and standard deviations of those signal intensities relative to the averaged signal noise per subject are the prime outcomes

SECONDARY OUTCOMES:
healthy-cohort signal resolution and uncertainty characteristics for metabolites of interest (MOI) | 2 months
  cohort characteristics of the resolution parameters (full width at half maximum intensity) and (where a fitting model is available) the uncertainties of the model fit from single subjects

CONTACTS AND LOCATIONS:
Overall Officials: Roland Kreis, PhD, Principal Investigator — Inselspital Bern & University Bern
Locations (1):
- Translational Imaging Center, Bern, PhD, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: project description on funders portal — https://p3.snf.ch/Project-175984